CLINICAL TRIAL: NCT00286611
Title: Serial Blood and Salivary Sampling for Validation of Quantitative Amifostine Assays
Brief Title: Determination of Amifostine Levels During Radiation Therapy
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: John Buatti, M.D., Department of Radiation Oncology
Other Study IDs: 200406002
Record Dates: First submitted 2006-01-31; First posted 2006-02-03 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Cancer
Keywords: Amifostine
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Amifostine: Those individuals enrolled who have received amifostine as part of standard care.
  Interventions: Procedure: Blood and salivary sampling of amifostine

INTERVENTIONS:
Procedure: Blood and salivary sampling of amifostine — Sampling of blood and saliva to test for amifostine levels.

SUMMARY:
Currently, there are no published methods for easily determining the level of amifostine in the blood or saliva. A method has been developed within the Department of Radiation Oncology by Drs. Douglas Spitz and Gurminder Sidhu, within the Spitz Lab. This method has been tested using both animal sampling and expired blood (obtained from DeGowin blood center) mixed with amifostine.

If the method proves successful, it could then be used as a tool to quantify blood and salivary amifostine levels and possibly correlate them to treatment efficacy or limiting adverse events using amifostine. A better method of treatment, either increasing the efficacy of amifostine or reducing its unwanted side effects, could then be developed.

DETAILED DESCRIPTION:
Currently, there are no published methods for easily determining the level of amifostine in the blood or saliva. A method has been developed within the Department of Radiation Oncology by Drs. Douglas Spitz and Gurminder Sidhu, within the Spitz Lab. This method has been tested using both animal sampling and expired blood (obtained from DeGowin blood center) mixed with amifostine.

If the method proves successful, it could then be used as a tool to quantify blood and salivary amifostine levels and possibly correlate them to treatment efficacy or limiting adverse events using amifostine. A better method of treatment, either increasing the efficacy of amifostine or reducing its unwanted side effects, could then be developed.

Amifostine is an FDA-approved medication that protects the lining of the mucous membranes of the head and neck when radiation treatments are given. Normally, amifostine is injected into a vein causing side effects of nausea, vomiting and low blood pressure. The amifostine can reduce radiation side effects but does not remove them completely.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent document.
* Receiving radiation treatment at University of Iowa Hospitals and Clinics.
* Voluntarily elected to receive amifostine during treatment

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients receiving amifostine as a part of their standard cancer therapy.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2004-10; Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. Buatti, M.D., Principal Investigator — University of Iowa Hospitals & Clinics; Douglas R. Spitz, Ph.D., Study Director — Carver College of Medicine University of Iowa
Locations (1):
- University of Iowa Department of Radiation Oncology, Iowa City, Iowa, United States